CLINICAL TRIAL: NCT02989311
Title: Testing Iron Absorption From a New Micronutrient Powder Containing Galacto-oligosaccharides (GOS) for Fortification of Infant Foods in Sub-Saharan Africa
Brief Title: Effect of Timing of Micronutrient Powder Consumption on Iron Absorption in Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: Jomo Kenyatta University of Agriculture and Technology (Other); Msambweni County Referral Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: FeGOS_Hepcidin
Record Dates: First submitted 2016-10-18; First posted 2016-12-12 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2016-12

CONDITIONS: Anemia; Iron Deficiency
Keywords: Iron absorption; Iron deficiency; Hepcidin; Stable isotopes; Anemia; Infants
MeSH Terms: conditions — Anemia; Iron Deficiencies | interventions — Iron

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Study 1:Morning test meal+Iron+MNP (Active Comparator): The MNP contains 400 μg Vitamin A, 5 μg Vitamin D, 5 mg Tocopherol Equivalent, 0.5 mg Thiamine, 0.5 mg Riboflavin, 0.5 mg Vitamin B6 , 90 μg Folic Acid,6 mg Niacin, 0.9 μg Vitamin B12, 30 mg Vitamin C, 0.56 mg Copper, 90 μg, Iodine, 17 μg Selenium, 4.1 mg Zinc, 190 Phytase-units, plus 2.5 mg Fe as Ferrous Fumarate and 2.5 mg Fe as NaFeEDTA, maltodextrin carrier (added up to 11g). Iron compound added to the morning test meal A:12 mg of iron as ferrous sulfate given as 2 mg of 57Fe and 10mg of 56Fe.
  Intervention: Dietary supplement: Fortified maize porridge (MNP + Iron)
  Interventions: Dietary Supplement: Fortified maize porridge (MNP and Iron)
- Study 1:Afternoon test meal+Iron+MNP (Active Comparator): The MNP contains 400 μg Vitamin A, 5 μg Vitamin D, 5 mg Tocopherol Equivalent, 0.5 mg Thiamine, 0.5 mg Riboflavin, 0.5 mg Vitamin B6 , 90 μg Folic Acid,6 mg Niacin, 0.9 μg Vitamin B12, 30 mg Vitamin C, 0.56 mg Copper, 90 μg, Iodine, 17 μg Selenium, 4.1 mg Zinc, 190 Phytase-units, plus 2.5 mg Fe as Ferrous Fumarate and 2.5 mg Fe as NaFeEDTA, maltodextrin carrier (added up to 11g). Iron compound added to the afternoon test meal B:12 mg of iron as ferrous sulfate given as 2 mg of 58Fe and 10mg of 56Fe.
  Intervention: Dietary supplement: Fortified maize porridge (MNP + Iron)
  Interventions: Dietary Supplement: Fortified maize porridge (MNP and Iron)
- Study 2: Consecutive meals+Iron+MNP+GOS (Active Comparator): The MNP contains 400 μg Vitamin A, 5 μg Vitamin D, 5 mg Tocopherol Equivalent, 0.5 mg Thiamine, 0.5 mg Riboflavin, 0.5 mg Vitamin B6 , 90 μg Folic Acid,6 mg Niacin, 0.9 μg Vitamin B12, 30 mg Vitamin C, 0.56 mg Copper, 90 μg, Iodine, 17 μg Selenium, 4.1 mg Zinc, 190 Phytase-units, plus 2.5 mg Fe as Ferrous Fumarate and 2.5 mg Fe as NaFeEDTA, plus 7.5 g of galacto-oligosaccharides given as 10.5 g GOS-75, maltodextrin carrier (added up to 11g) Iron compound added to the test meals:Test meal A will contain 12mg of ferrous sulphate given as 2mg 54Fe and 10mg 56Fe. Test meal B will contain 12mg of ferrous sulphate given as 2mg 57Fe and 10mg 56Fe.
  Intervention: Dietary supplement: Fortified maize porridge (MNP+ Iron + GOS)
  Interventions: Dietary Supplement: Fortified Maize porridge (MNP + Iron + GOS)
- Study 2:Alternate meal+Iron+MNP+GOS (Active Comparator): The MNP contains 400 μg Vitamin A, 5 μg Vitamin D, 5 mg Tocopherol Equivalent, 0.5 mg Thiamine, 0.5 mg Riboflavin, 0.5 mg Vitamin B6 , 90 μg Folic Acid,6 mg Niacin, 0.9 μg Vitamin B12, 30 mg Vitamin C, 0.56 mg Copper, 90 μg, Iodine, 17 μg Selenium, 4.1 mg Zinc, 190 Phytase-units, plus 2.5 mg Fe as Ferrous fumarate and 2.5 mg Fe as NaFeEDTA, plus 7.5 g of galacto-oligosaccharides given as 10.5 g GOS-75, maltodextrin carrier (added up to 11g) Iron compound added to the test meal C: 12mg of ferrous sulphate given as 2mg 58Fe and 10mg.
  Intervention: Dietary supplement: Fortified maize porridge (MNP+ Iron + GOS)
  Interventions: Dietary Supplement: Fortified Maize porridge (MNP + Iron + GOS)

INTERVENTIONS:
Dietary Supplement: Fortified maize porridge (MNP and Iron) — Maize porridge fortified with MNP and labelled iron compound
  Arms: Study 1:Afternoon test meal+Iron+MNP; Study 1:Morning test meal+Iron+MNP
Dietary Supplement: Fortified Maize porridge (MNP + Iron + GOS) — Maize porridge fortified with MNP + GOS and labelled iron compound
  Arms: Study 2: Consecutive meals+Iron+MNP+GOS; Study 2:Alternate meal+Iron+MNP+GOS

SUMMARY:
Infants and young children in sub-Saharan Africa have high rates of iron deficiency anemia (IDA), which adversely affects their growth and cognitive development. In-home iron fortification of complementary foods using micronutrient powders (MNPs) reduces risk for IDA by ensuring that the iron needs of infants and young children are met without changing their traditional diet. In order to optimize iron absorption timing of MNP consumption might as well be important. This is because hepcidin, a key regulator of systemic iron balance, shows a circadian increase that may influence morning versus afternoon iron absorption from the MNP. Furthermore, a single dose of iron can increase hepcidin levels and potentially inhibit iron absorption from a second dose, consumed close in time to the first dose.

To determine the difference between i) morning versus afternoon iron absorption and ii) consecutive versus alternate day iron absorption, investigators will enrol 20 infants from Kwale County aged 6-14 months and conduct two studies. In study 1, infants will consume 2 test meals consisting of maize porridge containing isotopically labelled Ferrous Sulphate in the morning and afternoon on 2 days. In study 2, infants will consume 3 test meals consisting of maize porridge containing isotopically labelled Ferrous Sulphate on two consecutive days and 1 alternate day. In both studies, fourteen days after the last test meal administration, a whole blood sample will be collected by venipuncture for iron isotopic analysis. Iron and inflammation status parameter will be determined at baseline and endpoint. Hepcidin concentrations will be measured before the morning and afternoon meals (study 1) and after second consecutive meal (study 2).

Knowing the effect of time on the expected iron absorption will inform decisions on the ideal timing of MNP to cover the infant's requirement for absorbed iron.

DETAILED DESCRIPTION:
20 infants will be recruited from the Msambweni County Referral Hospital in southern coastal Kenya to participate in both studies.

Study 1:

At baseline a morning blood sample will be collected from potential study participants for the determination of the following iron and inflammation status parameters: hemoglobin (Hb), hepcidin, plasma ferritin (PF), soluble transferrin receptor (sTfR), zinc protoporphyrin (ZnPP), C-reactive protein (CRP), alpha-1-acid glycoprotein (AGP). Anthropometrics (height, weight, mid-upper arm and head circumference) will be measured, and demographics, the medical history and the feeding habits will be assessed using a questionnaire.

Infants will consume the 1st test meal the next day after enrolment in the morning (day1). On day 2 a 2nd blood sample (1ml) will be collected in the afternoon quantify afternoon concentration of hepcidin in plasma and then the infants will consume the 2nd meal on the 3rd day in the afternoon.

The two isotopically labelled test meals will be fed to the infants by their caregivers under supervision of the research team. The morning test meal A will contain 12 mg of iron as ferrous sulfate given as 2 mg of 57Fe and 10mg of 56Fe. The afternoon test meal will contain 12 mg of iron as ferrous sulfate given as 2 mg of 58Fe and 10 mg of 56Fe.

The test meals will consist of maize porridge (5-10% dry weight) and mineral water (8ml) and will be randomly administered on the two alternate days (AB or BA). Overnight, only breast milk will be allowed to the infant before coming for the morning meal and no breast milk will be given at least 3 h before both morning and afternoon test meal administration. Infants will not be allowed to eat or drink for 2 h after the test meal. Fourteen days after the second test meal administration, 3 ml of whole blood will be collected by venipuncture for iron isotopic analysis and iron and inflammation status. Anthropometrics and health status will be assessed.

Study 2:

At baseline a blood sample will be collected from potential study participants for the determination of iron and inflammation status parameters: hemoglobin (Hb), hepcidin, plasma ferritin (PF), soluble transferrin receptor (sTfR), zinc protoporphyrin (ZnPP), C-reactive protein (CRP), alpha-1-acid glycoprotein (AGP). Anthropometrics (height, weight, mid-upper arm and head circumference) will be measured, and demographics, the medical history and the feeding habits will be assessed using a questionnaire.

Infants will be randomized to consume the consecutive days or alternate day meal schedule on day 1. 1ml of blood will be collected after the second consecutive meal to determine hepcidin level.

Test meal A will contain 12 mg of iron as ferrous sulfate given as 2 mg of 54Fe and 10mg of 56Fe. Test meal B will contain 12 mg of iron as ferrous sulfate given as 2 mg of 57Fe and 10mg of 56Fe. Test meal C will contain 12 mg of iron as ferrous sulfate given as 2 mg of 58Fe and 10mg of 56Fe. All test meals will be consumed in the morning.

The test meals will consist of maize porridge (5-10% dry weight) and mineral water (8ml). Overnight, only breast milk will be allowed to the infant and no breast milk will be given at least 3 h before test meal administration. Test meals plus mineral water will be consumed completely in the presence of the investigators, and the infant will not be allowed to eat or drink for 2 h after the test meal. Fourteen days after the third test meal, 3 ml of whole blood will be collected by venipuncture for iron and inflammation status, and iron analysis in red blood cells.

ELIGIBILITY:
Inclusion Criteria:

* Age of 6-14 months at baseline
* Assessment of good health as assessed by health professional staff at Msambweni County Referral Hospital
* Willingness of their caregiver to provide informed consent

Exclusion Criteria:

* Hemoglobin <70 g/L; these infants will be referred for treatment according to local standard of care
* Severe underweight (Z-score weight-for-age <-3) and /or severe wasting (Z-score weight-for-height<-3)
* Chronic or acute illness or other conditions that in the opinion of the Principle Investigator (PI) or co-researchers would jeopardize the safety or rights of a participant in the trial or would render the participant unable to comply with the protocol
* Participants taking part in other studies requiring the drawing of blood
* Participants who are taking iron-containing food supplements or tablets/drops

Ages: 6 Months to 14 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2016-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in isotopic ratio of iron in blood at day 18 and 19 for Study 1 and 2 respectively | Baseline and day 18, baseline and day 19

SECONDARY OUTCOMES:
Hepcidin concentration | Baseline and day 3, and day 2 for study 1 and 2 respectively
  We will measure hepcidin concentration in the morning and in the afternoon and then after consumption of a 2nd consecutive test meal in Study 1 and 2 respectively
Iron status | Baseline and days 18 and 19 for study 1 and 2 respectively
  We will assess haemoglobin, plasma ferritin and soluble transferrin receptor to define the iron status.
Inflammation status | Baseline and days 18 and 19 for study 1 and 2 respectively
  We will assess C-reactive protein and alpha acid glycoprotein to assess systemic inflammatory status

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zimmermann, MD, Principal Investigator — Swiss Federal Institute of Technology (ETH), Zurich
Locations (1):
- Msambweni County Referral Hospital, Msambweni, Kwale County, Kenya

IPD SHARING:
Plan to Share IPD: Yes
Data will be published in a peer-review journal

REFERENCES:
- [Derived] Uyoga MA, Mikulic N, Paganini D, Mwasi E, Stoffel NU, Zeder C, Karanja S, Zimmermann MB. The effect of iron dosing schedules on plasma hepcidin and iron absorption in Kenyan infants. Am J Clin Nutr. 2020 Oct 1;112(4):1132-1141. doi: 10.1093/ajcn/nqaa174. PMID 32678434